CLINICAL TRIAL: NCT03085030
Title: Effect of Some Antioxidants on the Conception Rate in Poor Responders in IVF Cycles (a Randomized Controlled Trial)
Brief Title: Can Antioxidants Affect Pregnancy Rate in Patients With Expected Low Number of Egg Retrieval in IVF Cycles?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Omran, lecturer and consultant of Obstetrics and Gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3656
Record Dates: First submitted 2017-03-15; First posted 2017-03-21 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Infertility, Female
Keywords: infertility; IVF; ICSI; poor responders in IVF/ICSI cycles; antioxidant
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Intervention Model Description: The first group will take antioxidant drug orally once daily for one month before IVF/ICSI cycle.
  The second group will take placebo with a same regimen as the antioxidant group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both the antioxidant and the placebo will be put in sealed envelops with a number on it. the number denotes its order in the randomization process. The investigator, care providers and the outcome assessors will not know the allocated group of the participants. The bio-statistician will prepare the table of random numbers. the pharmacist will prepare the sealed envelopes according to the table of randomization. Independent nurse will bring the sealed envelope of the participant from the pharmacy without knowing whether the envelope contains drug or the placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- antioxidant group (Experimental): This group will take antioxidant formula tablet once daily orally for one month before IVF/ICSI cycle
  Interventions: Drug: Antioxidant Formula
- control group (Placebo Comparator): This group will take placebo tablet once daily orally for one month before IVF/ICSI cycle
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Antioxidant Formula — Antioxidant tablet will be taken by the patients
  Arms: antioxidant group
Drug: Placebo — The placebo will be taken by the patients
  Arms: control group

SUMMARY:
The aim of the study is to evaluate the effect of antioxidants on IVF outcome in infertile patients undergoing IVF who are expected to produce low number of eggs compared to a control group. The investigators assumed that the conception rate is higher in those patients taking some antioxidants supplementation. The patients will be given antioxidant drug one month before starting IVF trial once daily by mouth. Uniform protocol of stimulation will be done during the cycle by a type of short protocols known as the antagonist protocol. Egg retrieval will be done under anesthesia. pregnancy test will be done 2 weeks after embryo transfer. The investigators will also assess the number and quality of eggs on the day of egg pick up. In addition, the researchers will assess the number of first and second grade embryos that are put on the day of embryo transfer.

DETAILED DESCRIPTION:
The primary aim of this study is to assess the value of antioxidant intake on the pregnancy rate in IVF/ICSI (invitro-fertilization/intracytoplasmic sperm injection) cycles in poor responders. when the participants fulfill the eligibility criteria, informed consent will be taken. Block randomization will be done and the patients are allocated to one of two groups. The first group will take the antioxidant tablet daily orally for one month before the IVF/ICSI cycle. the other group will take placebo following the same regimen as the study group. Antagonist protocol will be done for all participants. Ovum pick up will be done under general anesthesia when one or more oocytes reaches 17 mm. The researchers will do embryo transfer on day 2 or 3 after ovum pickup. pregnancy test will be in blood after 2 weeks of embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

Infertile females undergoing IVF/ICSI cycles Poor responders are identified with

1. A previous poor ovarian response (less than 3 oocytes with a conventional ovarian stimulation protocol)
2. An abnormal ovarian reserve test which is considered altered in case of antral follicle count less than 5 follicles or AMH (anti-mullerian hormone) less than 1.5 ng/ml.
3. FSH (follicle stimulating hormone) value more than 10 IU/mL .

Exclusion Criteria:

1. Any endocrine or metabolic disorders such as diabetes and thyroid dysfunction
2. Any significant uterine anomaly, uterine cavity distortion, fibroids, hydrosalpinx or advanced endometriosis of stage III to IV
3. Severe oligo-astheno-teratozoospermia or azoospermia are excluded, as well.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 593 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
pregnancy rate | pregnancy test will be done 2 weeks after the IVF/ICSI trial for each participant
  pregnancy rate in the antioxidant and placebo groups.

SECONDARY OUTCOMES:
The number oocytes retrieved | At the time of egg retrieval
  The number oocytes retrieved for each participant
number of good quality eggs | At the time of egg retrieval
  at the time of egg retrieval for each participant
number of grade 1 and 2 embryos | number of grade 1 and 2 embryos at time of embryo transfer
  number of grade 1 and 2 embryos for each participant

CONTACTS AND LOCATIONS:
Overall Officials: Eman F Omran, M.D., Principal Investigator — Cairo University
Locations (1):
- Department of Obstetrics and Gynecology, Kasr Al-Ainy hospital, Cairo, Greater Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No